CLINICAL TRIAL: NCT02628340
Title: Comprehensive Analysis of HIV Reservoirs in Chronically Infected HIV-1 Treated Patients With a Low Total Cell-associated Blood HIV-DNA
Brief Title: Comprehensive Analysis of HIV Reservoirs in Chronically Infected HIV-1 Treated Patients
Acronym: RESACHRON
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Collaborators: INSERM UMR S 1136 (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CREPATS 002
Record Dates: First submitted 2015-02-04; First posted 2015-12-11 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: HIV

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Ex-vivo analysis

SUMMARY:
HIV infection can be efficiently controlled by antiretroviral therapy (ART), with in 2013 nearly 85 % of patients having a suppressed viremia, but HIV cannot, however, be eradicated with ART alone [1]. Overall, HIV has moved from a fatal to a chronic disease provided treatment is maintained life-long. Despite major improvement in antiretroviral drugs in terms of efficacy, tolerability and simplicity, life-long therapy is still associated with drug toxicity. Several drugs or drug classes, which have historically saved lives since 1996 and are currently widely used such as protease inhibitors and nucleosides analogues, are associated with long-term toxicities and increased incidence of comorbidities.

Currently, worldwide there is an approximated 10 millions of HIV infected patients under cART. This number should increase in the next years, as most recent guidelines recommend earlier therapy given the benefits in terms of disease progression and prevention of transmission. Because of the increasing number of patients who will be under cART in the future, the cumulative ART toxicity, the difficulties to access ART in some areas of the world, the fatigue expressed by patients about ART and the cost issues, there is an urgent need to search for HIV CURE. To date, only two cases of sterilizing HIV cure were reported so far: the famous "Berlin Patient" after two homozygous Delta32-CCR5 bone-marrow grafts for an acute leukemia [2], and the Mississipi baby after very early initiation of cART 31 hours after delivery [3]. However those cases of sterilizing HIV cure remain exceptional and the alternative objective of a functional HIV cure appears to be more realistic, though still described in rare groups of patients like Elite controllers (EC) and post treatment controllers (PTC) patients. In addition new and complex therapeutic strategies are currently proposed to try purging the HIV reservoirs, but none of them proved so far able to reach this goal.

Therefore the objective of finding a Cure to HIV [4] requires first to better understand the basic mechanisms of the persistence of HIV reservoirs in the population of chronically-infected fully-suppressed HIV+ patients in order to define future therapeutic strategies.

DETAILED DESCRIPTION:
Extremely low levels of HIV reservoirs are achievable in some chronically-infected patients durably controlled with cART. Despite the multiplicity and heterogeneity of factors governing the persistence of HIV reservoirs, such low levels of HIV reservoirs seem necessary, though probably not sufficient, to reach the status of functional cure defined by virus control in the absence of treatment. The mechanisms associated with these low HIV reservoirs in chronic treated infection are unknown but might involve a low immune activation and inflammatory environment, and deleterious HIV mutations. Understanding those mechanisms will provide novel clues for future strategies aiming at obtaining an HIV Cure.

The main objective of RESACHRON Study is to define in chronically infected patients with suppressed viremia, cART and extremely low levels of HIV reservoirs, the viral and cellular mechanisms underlying the persistence, the size and the distribution of these HIV reservoirs among the various CD4 T cell-subpopulations via a comprehensive analysis using innovative highly miniaturized and complementary immunological and virological assays.

Our first hypothesis is that HIV reservoirs persist even in patients with low to undetectable HIV-DNA in the total PBMCs, and can be detected ex vivo or give rise to HIV production in some CD4 T cells subsets due to the mean 10-fold enrichment in peripheral blood TCM and TTM cells. The sorting of the various sorted CD4 TN, TCM, TTM, TEM and other key subsets will thus allow to test whether and in which subset:

1. the virus genome is intact or contains deletions interfering with its replicative capacity,
2. HIV production can be induced in vitro after distinct activation signals,
3. HIV transcripts are detectable ex-vivo,
4. Low immune activation and inflammatory environment is associated with these extremely low HIV reservoirs levels by testing a series of plasma pro-inflammatory molecules together with cell surface activation markers and intra-cellular transcriptional signatures .

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adult
* Age > 18 years
* HIV-RNA plasma viral load (pVL) < 50 copies/mL
* Under antiretroviral therapy (cART)
* CD4 >400/mm3
* HIV DNA<200 copies/106 PBMCs
* Ability to provide informed consent

Exclusion Criteria:

* cART initiated at the time of primary infection
* Chronic hepatitis B ( HBs +antigen)
* Chronic hepatitis C defined as positive HCV-RNA
* History of chemotherapy/radiotherapy or immunosuppressive therapy within the 5 years prior study entry.
* Any history of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 patients under cART with HIV-RNA pVL < 50 cp/ml and HIV DNA <200 copies/106 PBMCs will be recruited from a total of over 3,900 patients under follow-up in the Infectious Diseases Unit Pitié-Salpêtrière Hospital, in Paris.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
measure of HIV reservoirs in a selected HIV chronically infected ARV treated population assessed by HIV DNA distribution in PBMCs, total and sorted CD4 T cells subsets. | one year
  Cell sorting experiments will allow the sorting of the different subsets of the CD4 reservoirs cells and their quantification for the study of the HIV reservoirs characteristics. We will sort resting CD4 T cells defined as CD3+CD4+CD69-CD25-HLA-DR- on a 5-laser flow cytometer in our L3 facility (UPMC Platform CyPS) in at least 4 subsets:
  * Naïve (TN: CD45RA+CCR7+CD27+),
  * Central-Memory (TCM: CD45RA-CCR7+CD27+),
  * Transitional-memory (TTM: CD45RA-CCR7-CD27+)
  * Effector-Memory (TEM CD45RA-CCR7-CD27-)

SECONDARY OUTCOMES:
measure of host molecular signatures and transcriptional activity in each subset assessed by microfluidic qRT-PCR (Fluidigm) | one year
  host molecular signatures and transcriptional activity performed by using microfluidic qRT-PCR (Fluidigm) quantifying the key host's genes among a panel of 90 host's molecular signatures including factors involved in restriction, repression or activation of HIV transcription
measure of in vitro inducibility of the HIV provirus in the different sorted CD4 subsets harboring the HIV réservoirs assessed by ultrasensitive real-time RT-PCR assay | one year
  The induction of replication-competent HIV forms measured in culture supernatants from each subset by using the ultrasensitive real-time RT-PCR assay
measure of defective viral population estimated by the proportion of stop codons in the integrated HIV-DNA assessed by ultra deep sequencing and | one year
  ex vivo molecular characteristics phylogenetic analysis of the integrated HIV-DNA in the genome of sorted host CD4 subsets
measure of levels of unspliced HIV transcripts in total and different subsets of CD4 T cells. | one year
  Levels of unspliced HIV transcripts performed by using microfluidic qRT-PCR (Fluidigm)
measure of serum inflammatory biomarkers assessed by ELISA assay | one year
  Inflammatory biomarkers analyzed on plasma: hsCRP, IL6, sTNF I, IP-10, sCD14, sCD63 and D-dimers
measure of immune activation in the different sorted CD4 T cell subsets assessed by flow cytometry on fresh blood | one year
  • The cell immune activation markers analyzed by flow cytometry on fresh blood. Activation markers will be analyzed on CD4 (HLA-DR) and CD8 (HLA-DR, CD38) subsets (ie N, TCM, TTM, TEM) and on monocytes subsets defined by the expression of CD14/CD16 (CD163/CD38). The expression of CD38 will be quantified by beads.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Study Director — Groupe Hospitalier Pitié-Salpêtrière; Ruxandra Calin, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière - Service des Maladies Infectieuses et Tropicales, Paris, France